CLINICAL TRIAL: NCT02346500
Title: Ultrasound-Guided Photoselective Vaporization of the Prostate
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00052503
Record Dates: First submitted 2013-10-28; First posted 2015-01-27 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; Lower urinary tract symptoms; Photoselective laser vaporization of the prostate; Transrectal Ultrasound
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Ultrasound, High-Intensity Focused, Transrectal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transrectal ultrasound (Experimental): TRUS and TRUS-Robot will be used during PVP
  Interventions: Device: Transrectal Ultrasound

INTERVENTIONS:
Device: Transrectal Ultrasound — The TRUS and TRUS-Robot will be used to record ultrasound images during PVP. The PVP procedure will be conducted as usual, without using the ultrasound for guiding the intervention.

SUMMARY:
Benign prostatic hyperplasia (BPH) is a major cause of lower urinary tract symptoms (LUTS) affecting aging men. Medical therapy for BPH includes alpha adrenergic blockers and 5α-reductase inhibitors. In men with moderate-severe LUTS due to BPH, surgical therapy should be considered for 1) those who failed medical therapy and/or 2) those with refractory urinary retention, renal insufficiency secondary to BPH, recurrent urinary tract infections (UTI's), or bladder stones. The gold standard for the surgical therapy of BPH has been transurethral resection of the prostate (TURP). However, TURP is associated with significant comorbidities such as bleeding, prolonged catheterization, and absorptional hyponatremia. To minimize these problems associate with TURP, alternative minimally invasive treatment techniques have been developed. Two of the most commonly used treatment modalities include a photoselective laser vaporization of the prostate (GreenLight PVP) using the potassium titanyl phosphate (KTP) laser and holmium laser enucleation of prostate (HoLEP). The major problem in all these minimally invasive treatment modalities is that they are generally associated with a higher retreatment rate. In addition, there is no intraoperative and objective measurement, other than a limited, transurethral visualization of the prostatic cavity, to assess the extent of the vaporization or enucleation.

We propose to use the transrectal ultrasound (TRUS) and a novel robot, the TRUS robot, to hold and manipulate the TRUS probe to monitor the extent of the vaporization or enucleation of the prostate gland intraoperatively. TRUS has been extensively used for the biopsy needle guidance during prostate biopsy. However, it has never been used during transurethral prostate procedure. The TRUS Robot has been used safely in the current clinical trial, NA_00027540, Ultrasound-Guided Navigation in Robot-Assisted Laparoscopic Radical Prostatectomy. We would like to study the feasibility and safety of using TRUS and the TRUS Robot to monitor the minimally invasive treatment of BPH, such as GreenLight PVP.

DETAILED DESCRIPTION:
In the current pilot safety and feasibility (S&F) study for ultrasound-guided PVP (UG-PVP), we propose to use TRUS and the TRUS-Robot to record ultrasound images during PVP in 10 patients. The PVP procedure will be conducted as usual, without using the ultrasound for guiding the intervention. TRUS images of the prostate gland and the intraprostatic cavity formed during the PVP procedure will be recorded. These will include three dimensional (3-D) images acquired at the beginning and end of the operation. In addition, real-time 2-D images will be recorded during the case. Recorded images will then be analyzed offline to observe the extent of the vaporization or enucleation of the prostate gland.

ELIGIBILITY:
Inclusion Criteria:

* patients between the ages of 40 and 85
* patients with BPH
* patients scheduled for PVP

Exclusion Criteria:

* patients with known prostate cancer
* patients with bleeding problems
* patients with previous rectal surgery
* patients with anal stenosis
* patients who cannot tolerate anesthesia or in whom anesthesia is considered high-risk
* patients with previous pelvic irradiation
* patients with penile implants
* patients with artificial urinary or rectal sphincters
* patients who are unwilling or unable to sign informed consent

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2016-11-26 (Actual); Study Completion 2016-11-26 (Actual)

PRIMARY OUTCOMES:
Measurement of prostate volume. | During the study procedure, after the TRUS probe is in position for imaging of the prostate.
  Prostate volume will be measured before (Set I, initial: 3 min) and after (Set F, final: 3 min) the PVP.
Measurement of the prostate cavity. | At the end of the PVP procedure.
  Measurement will be estimated from the 3-D ultrasound Set F.
Recording patient-completed questionnaires (International Prostate Symptom Score (IPSS). | Measurements will be recorded 3 months after the PVP procedure.

SECONDARY OUTCOMES:
Measurement of complications from the procedure including rectal injury. | Measurements will be recorded during the PVP procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Misop Han, M.D., M.S., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States